CLINICAL TRIAL: NCT05391035
Title: The Antibiotic Guardian Study- a Clinical Evaluation of a Rapid Diagnostic of Mycoplasma and Gonorrhoea Infections and Antibiotic Resistance.
Brief Title: The Antibiotic Guardian Study- Clinical Evaluation of a Novel, Rapid Diagnostic for Gonorrhoea and Mycoplasma Infections.
Acronym: Guardian
Status: Completed | Type: Observational
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: CT 269508
Record Dates: First submitted 2021-12-23; First posted 2022-05-25 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2021-11

CONDITIONS: Sexually Transmitted Diseases, Bacterial; Antibiotic Resistant Infection
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic patients attending a sexual health clinic.: A cohort of 160 symptomatic people attending a sexual health clinic in the UK will be recruited to this observational study.

SUMMARY:
Primary research question:

Are novel molecular tests for rapid detection of Mycoplasma and Gonorrhoea infections and antimicrobial resistance sensitive and specific in symptomatic patients attending a sexual health clinic?

Secondary research question:

Are novel molecular tests for detection of antimicrobial resistance in Mycoplasma and Gonorrhoea infections more accurate than standard laboratory culture techniques?

DETAILED DESCRIPTION:
This clinical study aims to clinically evaluate a novel, rapid molecular diagnostic for Mycoplasma and Gonorrhoea infections. This diagnostic detects both infection and also detects any antimicrobial resistance. These tests detect these organisms and provide information about antimicrobial resistance in a laboratory, but are not widely used in sexual health clinics in the UK and have not been clinically evaluated in symptomatic patients in detail.

Our primary objective is to determine if the novel molecular test for rapid detection of Mycoplasma and Gonorrhoea infections and antimicrobial resistance is sensitive and specific in symptomatic patients attending a sexual health clinic.

Our secondary research objective is to determine whether the novel molecular test for detection of antimicrobial resistance in Mycoplasma and Gonorrhoea infections more accurate than standard laboratory culture techniques.

Eligible participants will be aged between 16 and 99 years and attend a sexual health clinic at Cwm Taf Morgannwg Sexual Health department. They will be symptomatic.

Participants will have routine swabs performed as per routine sexual health care, following gaining participant consent in writing. Waste urine and discharge from vaginal swabs will be utilised in the study. Samples will be given a unique study number and sent to the normal NHS laboratory for analysis as per routine care. Left-over samples of urine and swabs will be pseudo-anonymised and then transported to the academic laboratory for analysis with the novel diagnostic with the unique study ID.

Results from routine tests for Mycoplasma and Gonorrhoea detection and for antimicrobial resistance will be compared to results of the novel diagnostic.

This study has had a substantial amendment reviewed and passed by an ethics committee, due to COVID disruptions in healthcare. It has changed from an interventional study to an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are sexually active.
* Patients that are symptomatic with:
* Dysuria
* Urethral discharge
* Vaginal discharge
* Rectal discharge
* Dysparenia (pain during sex)
* Pelvic pain
* Testicular pain
* Post-coital bleeding (bleeding after sex)
* Vulval/Glans/Perianal pain.

Exclusion Criteria:

* Pregnancy.
* Aged under 16 years.
* Sexual assault case.
* Patients with very severe symptoms that need admission to a ward or referral for urgent gynaecology or urology interventions.
* Patients lacking capacity to consent.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Symptomatic patients attending a sexual health clinic in Cwm Taf Morgannwg health board, UK.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of a novel, rapid diagnostic for the detection of Mycoplasma and Gonorrhoea | 3 years
  Investigators will determine the specificity and sensitivity of the novel molecular diagnostic in the detection of Mycoplasma and Gonorrhoea infections from clinical samples performed during testing of symptomatic participants. Results of the novel diagnostic will be compared to standard current laboratory test results and the results of quantitative PCR.

SECONDARY OUTCOMES:
Comparison of molecular tests and routine culture techniques for detection of antibiotic resistance in Gonorrhoea and Mycoplasma infections. | 3 years
  Investigators will determine the specificity and sensitivity of the novel molecular diagnostic in the detection of antimicrobial resistance in Mycoplasma and Gonorrhoea infections from clinical samples performed during testing of symptomatic participants. Results of the novel diagnostic will be compared to standard current laboratory test results for antibiotic resistance and and the results of sequencing Gonorrhoea and Mycoplasma bacteria for antibiotic resistance genes.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Cwm Taf Morgannwg University Health board, Llantrisant, Rhondda Cynon Taf
  - Lucy Jones, Pontypridd

IPD SHARING:
Plan to Share IPD: No
no plan to share participant data